CLINICAL TRIAL: NCT04021004
Title: How do Pilates Trained Physiotherapists Utilise and Value Pilates Exercise for MSK Conditions: A Qualitative Study
Status: Completed | Type: Observational
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Peter Cuddy, Postgraduate Student of Masters In Advanced Physiotherapy, University of Salford
Other Study IDs: Ref HSR1617-150
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: MSK Conditions
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey Questionnaire — Survey Questionnaire

SUMMARY:
A self-designed qualitative questionnaire survey was used to investigate opinions and views among thirty Physiotherapists practising in the UK, who had undertaken formal training in Pilates exercise therapy to treat people with MSK conditions.

DETAILED DESCRIPTION:
Pilates is a popular exercise therapy approach that focuses on strength, core stability, flexibility, muscle control, and posture (Wells et al., 2014). This approach has evolved over time, to form a valuable therapeutic tool in the prevention and rehabilitation of a variety of injuries (Di Lorenzo, 2011). More recently, Pilates has become increasingly popular due to its wide-ranging health benefits for individuals with a range of MSK (musculoskeletal) disorders, as well as other conditions (Byrnes, Wu, & Whillier, 2018). This method has become more commercially recognised and accessible through various professional institutions. The Australian Physiotherapy & Pilates Institute (APPI), is a globally run organisation licensed in sixteen countries, delivering over 17000 classes per year, as a "graduated system of specific exercise rehabilitation" (Appihealthgroup.com, 2018).

In the UK, Pilates based exercise therapy is used within both the National Health Service (NHS) and private healthcare sectors in the management of low back pain (LBP), general MSK pain, and various degenerative conditions (Yamato et al. 2015). An estimated 17.8 million people live with a musculoskeletal condition in the UK, around 28.9% of the total population (Global Burden of Disease network, 2016). Over 8.75 million people aged 45 and over have sought treatment for osteoarthritis (Arthritis Research UK, 2013), for which the main management strategy is exercise-based therapy. MSK healthcare services are under increasing pressure to provide care to the ageing population, and tackle the healthcare impact associated with inactivity (Hubbard et al., 2004). Group based exercise such as class Pilates, offers an accessible opportunity to increase activity levels in such individuals (Karlsson, Gerdle, Takala, Andersson, & Larsson, 2018).

There is considerable evidence that Pilates has numerous physical benefits and may improve self-management of MSK conditions. This includes a wealth of quantitative research, several systematic reviews have demonstrated positive improvements on pain, quality of life and functionality (Aladro-Gonzalvo, Araya-Vargas, Machado-Díaz, & Salazar-Rojas, 2013; Byrnes et al., 2018). However, of the Randomised Controlled Trials (RCTs) reviewed, high levels of heterogeneity were reported, in terms of sample (sub-types of back pain), exercise selection, delivery and frequency of treatment.

In contrast to this, there is a dearth of qualitative research evaluating Pilates as a treatment approach, mostly focusing on LBP populations (Gaskell & Williams, 2018). These methods can be valuable to review the definition, scope and rationale of Pilates treatment methods used by Physiotherapists, to provide optimum rehabilitation. Use of a qualitative approach could also gain understanding of how Physiotherapists utilise Pilates for a range of conditions other than LBP (Wells et al., 2014). Therefore, this study aims to investigate the variation in Pilates delivery and why, and in line with previous qualitative studies, further explore the perceived benefits, risks and rationale for this exercise approach. This is the first study to review NHS and private physiotherapists in their use of Pilates group exercise.

ELIGIBILITY:
Inclusion Criteria:

* To participate in the study and complete the survey, it was specified that participants needed to:

  1. Have undertaken some form of formal Pilates instruction training, such as the Matwork Foundation Pilates courses with the APPI (Australian Physiotherapy and Pilates Institute) or BCP (Body Control Pilates, 2018). Physiotherapists did not have to be a fully certified instructor to participate in the study, however, they must have completed a minimum of one formal Pilates Instruction course. Participants were required to specify this in the demographics section of the survey.
  2. Be registered with the HCPC (Health and Care Professions council) to currently practice as a Physiotherapist without restriction in the UK. The reasoning for only surveying Physiotherapists is in keeping with the rationale of previous studies (Wells et al., 2014; Allen, 2014; Brennan and French, 2008). Who have advocated that including only Physiotherapists with formal Pilates training guarantees similar standards of practice of participants, as standards and qualification level may vary otherwise. Additionally, extending the survey to other practioners would make further comparisons challenging through data analysis.
  3. Be computer literate, have e-mail access, time to commit to completion of the survey, and ability to understand written English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UK Physiotherapists who have completed formal Pilates instruction training
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Survey Questionnaire | 5 months
  Self-designed electronic survey to capture Physiotherapists opinions and views. The survey was comprised of both multiple choice selections, and open-ended questions in order to allow free text input and generate narrative for thematic analysis.
  No scale questions were utilised in this questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Gaskell, MSc, Study Director — University of Salford
Locations (1):
- University of Salford, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuddy P, Gaskell L. "How do Pilates Trained Physiotherapists utilize and value Pilates Exercise for MSK conditions? A Qualitative Study". Musculoskeletal Care. 2020 Sep;18(3):315-329. doi: 10.1002/msc.1463. Epub 2020 Apr 6. PMID 32250561